CLINICAL TRIAL: NCT01337765
Title: A Phase Ib, Open-label, Multi-center, Dose-escalation and Expansion Study of an Orally Administered Combination of BEZ235 Plus MEK162 in Adult Patients With Selected Advanced Solid Tumors
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BEZ235 Plus MEK162 in Selected Advanced Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2103; 2011-000421-74 (EudraCT Number); C4211009 (Other: Pfizer)
Record Dates: First submitted 2011-04-02; First posted 2011-04-19 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Solid Tumor
Keywords: BEZ235,; MEK162; RAS RAF mutations,; triple negative breast cancer; pancreatic cancer,; NSCLC progressed on EGFR TKI; PI3K/mTOR inhibitor,; MEK inhibitor; Advanced and selected solid tumors
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Pancreatic Neoplasms | interventions — dactolisib; binimetinib

ARMS (1):
- BEZ235 + MEK162 (Experimental)
  Interventions: Drug: BEZ235 + MEK162

INTERVENTIONS:
Drug: BEZ235 + MEK162

SUMMARY:
This is an open label, dose finding, phase Ib clinical trial to determine the maximum tolerated dose (MTD) and/or RP2D of the orally administered PI3K/mTOR inhibitor BEZ235 in combination with the MEK1/2 inhibitor MEK162. This combination will be explored in patients with EGFR mutant NSCLC which has progressed on EGFR inhibitors and triple negative breast cancer, as well as pancreatic cancer, colorectal cancer, malignant melanoma, NSCLC, and other advanced solid tumors with KRAS, NRAS, and/or BRAF mutations. Dose escalation will be guided by a Bayesian logistic regression model with overdose control. At MTD or RP2D, two expansion arms will be opened in order to further assess safety and preliminary anti-tumor activity of the combination of BEZ235 and MEK162.

Study drugs will be administered orally on a continuous schedule, MEK162 bid and BEZ235 qd, a treatment cycle is defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

* histologically/cytologically confirmed, advanced non resectable solid tumors
* Measurable or non-measurable, but evaluable disease as determined by RECIST 1.0

Exclusion Criteria:

* Patients with primary CNS tumor or CNS tumor involvement
* Diabetes mellitus - Unacceptable ocular/retinal conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-07-08 (Actual); Primary Completion 2013-03-22 (Actual); Study Completion 2013-03-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | during Cycle 1 of treatment with BEZ235 and MEK162
  A complete treatment cycle is defined as 28 days of daily continuois treatment with study drug combination

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | from Cycle 1 Day 1 until treatment discontinuation
  A complete treatment cycle is defined as 28 days of daily continuois treatment with study drug combination
Overall response rate, duration of response, time to response and progression free survival | every 8 weeks of treatment
Time versus plasma concentration profiles of BEZ235 and MEK162 | during the first cycle of treatment
  A complete treatment cycle is defined as 28 days of daily continuois treatment with study drug combination
Treatment-induced PI3K and MEK/ERK pathway signaling inhibition and evidence of biological activity in tumor | during the first cycle of treatment and at disease progression
  A complete treatment cycle is defined as 28 days of daily continuois treatment with study drug combination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (2):
  - Massachusetts General Hospital Mass General 2, Boston, Massachusetts
  - University of Texas/MD Anderson Cancer Center MD Anderson PSC, Houston, Texas
- Pfizer Investigative Site, Parkville, Victoria, Australia
- Pfizer Investigative Site, Toronto, Ontario, Canada
- Pfizer Investigative Site, Villejuif, France
- Pfizer Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.